CLINICAL TRIAL: NCT02553863
Title: A Randomised Controlled Trial to Assess the Effectiveness and Cost-effectiveness of Acupuncture in the Management of Chemotherapy-induced Peripheral Neuropathy
Brief Title: The Effectiveness and Cost-effectiveness of Acupuncture in Managing Chemotherapy-induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other); Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Alex MOLASIOTIS, Head of School, School of Nursing, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12131801
Record Dates: First submitted 2015-09-08; First posted 2015-09-18 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: chemotherapy induced peripheral neuropathy; acupuncture; pain; cost-effectiveness
MeSH Terms: conditions — Pain | interventions — Acupuncture Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Acupuncture for 30min [twice weekly for 8 weeks]
  Interventions: Procedure: Acupuncture
- Control group (Other): Standard care
  Interventions: Procedure: Standard care

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture for 30min [twice weekly for 8 weeks]
  Arms: Intervention group
Procedure: Standard care — Standard care
  Arms: Control group

SUMMARY:
The purpose of this study is to determine whether a course of acupuncture is effective in the management of peripheral neuropathy related pain in patients receiving chemotherapy.

DETAILED DESCRIPTION:
Participants and settings:

- Patients with lung, breast, head & neck, colorectal or gynaecological cancer receiving taxanes or platinum-derivative chemotherapy experiencing CIPN after the end of cycle one will be the population of the study. The study will take place in a large cancer centre in the territory (Prince of Wales Hospital).

Recruitment:

- Potential subjects will be identified (through clinic lists and databases of patients who are undergoing treatment) and approached initially by the relevant clinical team and screening then undertaken by research staff. The trial will be run ethically, details of which process can be seen under additional material.

Randomisation:

- Patients will be allocated to a group through computer-generated randomisation to be done at the Prince of Wales clinical trials unit. Randomisation will consist of minimisation with a random element (stochastic minimisation), balancing for the treatment types (taxanes or platinum analogues received) at a ratio of 1:1 to the two groups.

Intervention:

- The acupuncture intervention is described below based on the STRICTA recommendations for reporting acupuncture trials. In the acupuncture group, patients will receive, in addition to standard care, a standardised 30-minute acupuncture session needling specific body points although there will be flexibility in case some points cannot be punctured (ie. in case of lymphoedema), and alternative points (as in routine practice) may be selected by the therapists using their discretion to maintain an equal dose of treatment to all patients. The points will be standardised according to the clinical manifestations of the subjects.

Standard care:

- The comparison arm will be a standard care control arm.

Study duration:

- Treatment duration will be 8 weeks. The duration of each patient's involvement in the study will be 20 weeks (5 months) with assessments at baseline, end of 8-week treatment, 14 weeks and 20 weeks. Based on available numbers in the study hospital, recruitment will be at 10 subjects/month, requiring 11 months for trial recruitment. Four months are assigned for trial set up, preparation and staff training, 5 months for follow-up of last patient recruited, and 4 months for data cleaning, analysis and report writing (=24 months study).

Outcome measures:

1. Functional status and Quality of Life [baseline, week 8, week 14, week 20 to assess changes from baseline over time]

   Primary outcome is assessment of Pain at 8-weeks (end of acupuncture treatment): Pain: 'worst pain during past week' will be measured using the Brief Pain Inventory which measures pain intensity and its interference with function.
2. Secondary outcomes:

   * The NCI-Common Toxicity Criteria (CTC) for Adverse Events will be completed at baseline and week 8 to assess change from baseline. This is a physician based grading system that includes criteria and definitions for quantifying and grading CIPN (both neurosensory and neuromotor components). This grading scale comprises a sensory and motor assessment and utilises a 5-point scale ranging from grade 1 to grade 5. Previous studies demonstrated that the CTC scale is a quick to use, easy to administer and most useful in carrying out a screening procedure for choosing which patients need a neurological examination.
   * The Total Neuropathy Score clinical version (TNSc) will be completed at baseline and week 8 to assess change from baseline.. The TNS combines information obtained from grading of symptoms, signs, nerve conduction studies, and quantitative sensory tests, and provides a single measure to quantify neuropathy.
   * Functional assessment of cancer therapy (FACT/GOG-Ntx) will be completed at baseline, week 8, week 14, week 20 to assess changes from baseline over time. This is a 38-item self reported questionnaire, divided into two sub-scales: the first one is a 27-item general assessment of quality of life sub-scale (FACT-G) while the second one is a 11-item neurotoxicity sub-scale. This tool demonstrated good internal reliability and construct validity.
   * Consumption of analgesics will also be measured with a patient diary, as well as the presence of other related symptoms (ie. fatigue, sleep, etc) using the 10-item Symptom Distress Scale at baseline, week 8, week 14, week 20 to assess changes from baseline over time] .
3. Sensory examination [baseline and at the end of Acupuncture course -8 weeks- to assess change from baseline] Sensory examination will take place by the doctor/nurse using 10-g monofilament to lightly touch the patient's hands and feet bilaterally with the patients eyes closed. The monofilament test is a standardised plastic filament that will be pressed against parts of the hands and feet. When the filament bends, its tip is exerting a pressure of 10-gr. Abnormal responses including hyperesthesia, anesthesia or hypoesthesia will be recorded.

   * Neurophysiological testing will include a detailed motor nerve conduction study of the following nerves on the affected limbs. For upper limbs, the test will include: median nerve (bilateral) and ulnar nerve (bilateral). For lower limbs, the test will include peroneal nerve (bilateral), tibial nerve (bilateral). There will be provision of the most sensitive parameters to register any axonopathy or demyelination. Distal latencies, amplitudes and conduction velocities will be measured. F-waves will be also performed. For the sensory nerve conduction part, the following nerves will be studied. For upper limbs, the test will include: median nerve (bilateral) and ulnar nerve (bilateral). For lower limbs, it will include sural nerve (bilateral). We anticipate that the most common abnormalities will reside in the sensory nerve conduction study with axonal derangement as the most common manifestation. Knowing the test may cause a little bit discomfort to participants, so participation in the testing is voluntary. We expect that equal number of participants in the intervention group and control group will participate in the testing (n=25 per group).
   * Sociodemographic and treatment characteristics will be obtained from the patients' records or patients themselves at baseline. Patients will be asked about treatment expectations, how much they believe this method will help them alleviate their pain and how much faith they have in acupuncture (10-point scales). As CIPN is managed with dose reductions in clinical practice, chemotherapy dosage documentation (cumulative dosage received, dose reductions, dosage each cycle, completed number of cycles, chemotherapy type) will also be collected. The dosage information is necessary to use this data as a covariate in the data analysis, if the dosing is not constant across patients. Adverse effects will be monitored and collected from patients or researchers at each clinic visit for the duration of the acupuncture treatment.
4. Measurement of costs

We will explore the cost impact data and capture the frequency, type and extent of the costs of and service utilisation by patients. This will be done at week 14 only covering the period from start of treatment until week 14. This is the first time a cost evaluation is taking place in a cancer symptom-related acupuncture trial. More specifically, costs will be identified, measured and valued using a micro-costing approach (by which each component of resource use is identified, estimated and a unit cost derived from market prices and national estimates). The cost analysis will be performed from the perspective of the health service provider and from a societal perspective. Included in the health care provider costs will be those accrued by the hospitals and general practitioners. Costs to the patients and their families, including social care, will be considered as the additional costs for society. Indirect costs in terms of workdays lost will also included. Data will be collected prospectively and retrospectively using a questionnaire designed by the University of Leeds.multiple sources including patient records and patient self reported questionnaires. The questionnaires will determine health service utilisation as a result of CIPN (e.g. outpatient or general practitioner visits), patient out of pocket expenses such as over the counter medicines or transport together with use of services in the social sector such as home help and support from family and friends. Valuation of resource items including hospital resources (e.g. bed days and staff time) and community resources (e.g. general practitioner visits, home help) use will be carried out using national estimates; market prices will be assigned to medication; non-market items, specifically patient time and informal help provided by family and friends, will be valued using market wage rates; out of pocket expenses (e.g. bus fares) will also be obtained. We have used this approach successfully in a multisite acupressure trial with 500 patients

Data analysis:

- Analyses will include descriptive statistics to summarise the data, analysis of variance to assess between-groups differences for primary and each of the secondary outcomes, and regression analysis (such as ANCOVA) using the baseline pain score as covariate. 95% CIs will also be calculated. In more detail, while a t-test is adequate for analysis, analysis of covariance will be used with the baseline pain score as a covariate and centre and trial arm as grouping factors. Equivalent analyses will be performed for the week 20 data (although it is acknowledged that such analyses would not be independent of the 14-week scores, as it is likely the week-14 and week-20 values will be correlated). Drop-out cases and non-respondents will be asked to complete the primary outcome scale (1-item) and the 5 items of the CTC scale on CIPN in order to capture outcomes in as many patients as possible in the intention to treat analysis, and if this is not feasible, we will use data imputation (LVCF: last value carried forward). An intention-to-treat analysis will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of lung cancer receiving chemotherapy with curative intend, and breast or gynaecological cancer, head & neck and colorectal cancer stage I, II or III.
* Currently receiving neurotoxic chemotherapy (taxanes, cisplatin,,carboplatin, etc)
* Reporting tingling in hands/feet and other indications of chemotherapy-induced peripheral neuropathy (CIPN) after initiation of cancer treatments, confirmed to be indicative of CIPN by a consultant.
* Not using any medication for the prevention or treatment of CIPN for the past 31 months
* Willing to participate and be randomised to one of the study groups.
* No previously established peripheral neuropathy

Exclusion Criteria:

Exclusion criteria will include patients with needle phobia; Patients with low platelet count (<50,000); Comorbidity with a bleeding disorder; Pregnancy, or having received acupuncture treatment in the past three months. In addition, the ipsilateral arm of patients who have undergone axillary dissection will also be excluded from needling as well as lymphoedematous limbs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Pain | at baseline, end of 8-week treatment, 14 weeks and 20 weeks (the latter two to assess possible longer term effects)
  measured using the Brief Pain Inventory which measures pain intensity and its interference with function.

SECONDARY OUTCOMES:
Grade of CIPN | at baseline, end of 8-week treatment
  The NCI-Common Toxicity Criteria (CTC) for Adverse Events is a physician based grading system that includes criteria and definitions for quantifying and grading CIPN (both neurosensory and neuromotor components). This grading scale comprises a sensory and motor assessment and utilises a 5-point scale ranging from grade 1 to grade 5.
Severity of neuropathy | at baseline, end of 8-week treatment
  The Total Neuropathy Score clinical version (TNSc). The TNS combines information obtained from grading of symptoms, signs, nerve conduction studies, and quantitative sensory tests, and provides a single measure to quantify neuropathy
Quality of life | at baseline, end of 8-week treatment, 14 weeks and 20 weeks (the latter two to assess possible longer term effects)
  Functional assessment of cancer therapy (FACT/GOG-Ntx) is a 38-item self reported questionnaire, divided into two sub-scales: the first one is a 27-item general assessment of quality of life sub-scale (FACT-G) while the second one is a 11-item neurotoxicity sub-scale. This tool demonstrated good internal reliability and construct validity
Sensory examination | at baseline, end of 8-week treatment
  Sensory examination will take place by the doctor/nurse using 10-g monofilament to lightly touch the patient's hands and feet bilaterally with the patients eyes closed. The monofilament test is a standardised plastic filament that will be pressed against parts of the hands and feet. When the filament bends, its tip is exerting a pressure of 10-gr. Abnormal responses including hyperesthesia, anesthesia or hypoesthesia will be recorded.
Measurement of costs | at baseline, end of 8-week treatment, 14 weeks and 20 weeks (the latter two to assess possible longer term effects)
  We will explore the cost impact data and capture the frequency, type and extent of the costs of and service utilisation by patients. The cost analysis will be performed from the perspective of the health service provider and from a societal perspective. Included in the health care provider costs will be those accrued by the hospitals and general practitioners. Costs to the patients and their families, including social care, will be considered as the additional costs for society. Indirect costs in terms of workdays lost will also included. Data will be collected prospectively and retrospectively using a questionnaire designed by the University of Leeds.
Consumption of analgesics | at baseline, end of 8-week treatment, 14 weeks and 20 weeks (the latter two to assess possible longer term effects)
  Consumption of analgesics will also be measured with a patient diary, as well as the presence of other related symptoms (ie. fatigue, sleep, etc) using the 10-item Symptom Distress Scale
Motor nerve conduction | at baseline, end of 8-week treatment
  Neurophysiological testing will include a detailed motor nerve conduction study

CONTACTS AND LOCATIONS:
Overall Officials: Alex MOLASIOTIS, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin
  - Queen Elizabeth Hospital, Tsim Sha Tsui

REFERENCES:
- [Derived] Molassiotis A, Dawkins B, Longo R, Suen LK, Cheng HL, Mok T, Hulme CT, Yeo W. Economic evaluation alongside a randomised controlled trial to assess the effectiveness and cost-effectiveness of acupuncture in the management of chemotherapy-induced peripheral neuropathy. Acupunct Med. 2021 Feb;39(1):41-52. doi: 10.1177/0964528420920285. Epub 2020 May 13. PMID 32404001
- [Derived] Molassiotis A, Suen LKP, Cheng HL, Mok TSK, Lee SCY, Wang CH, Lee P, Leung H, Chan V, Lau TKH, Yeo W. A Randomized Assessor-Blinded Wait-List-Controlled Trial to Assess the Effectiveness of Acupuncture in the Management of Chemotherapy-Induced Peripheral Neuropathy. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419836501. doi: 10.1177/1534735419836501. PMID 30905173